CLINICAL TRIAL: NCT06221631
Title: Brain Aging - a Comparative Study in Healthy and Patients With Multiple Sclerosis as Model of a Chronic Neuroinflammatory Disorder (BrainAgeMS)
Brief Title: BrainAgeMS - a Comparative Study of Brain Aging in Healthy and Patients With Multiple Sclerosis
Acronym: BrainAgeMS
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Schweizerische Multiple Sklerose Gesellschaft (Other); University of Bern (Other)
Responsible Party: Principal Investigator, Alejandro León Betancourt, Medical Resident, Insel Gruppe AG, University Hospital Bern
Other Study IDs: ethic number 2023-D0110; 10001315 (Other: Swissmedic); CIV-23-12-045014 (Other: EUDAMED)
Record Dates: First submitted 2024-01-03; First posted 2024-01-24 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: Brain Aging; Multiple Sclerosis; Neurodegeneration; Quantitative MRI
MeSH Terms: conditions — Multiple Sclerosis; Nerve Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Healthy Controls: Healthy individuals with a predefined healthy lifestyle (s. inclusion/exclusion criteria), without any progressive disease or any neurological disorder (aside from primary headaches)
- Group 2: Patients with Multiple Sclerosis: Patients with MS with a similar healthy lifestyle (s. inclusion/exclusion criteria), who are able to walk without more than one-sided walking aid (max. EDSS of 6 points), no relapse activity in the last 6 months, without any other progressive disease or other neurological disorder (aside from primary headaches)

SUMMARY:
The purpose of this study is to investigate new quantitative MRI-sequences for assessment of age-specific data for the prediction of brain aging.

DETAILED DESCRIPTION:
After being informed about the study, healthy controls and patients with multiple sclerosis giving written informed consent will undergo blood examination (for determination of the biological age using the publicly available R-package algorithm BioAge), clinical examination (for motor, cognitive and psychological parameters) as well as an MRI-investigation with chemical exchange saturation transfer (CEST) and T1-relaxometry on a 7 Tesla MRI. Data from the healthy controls will be used to set up a normative brain age data set, that could be used for example to train a model for brain age prediction.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent signed by the subject

* Group 1: Any healthy individual between 18 and 65 years of age
* Group 2: Any individuals with any diagnosis of Multiple Sclerosis between 18 and 65 years of age and EDSS ≤6.0.

Exclusion Criteria:

* Group 1 and 2: Any other neurological disease except primary headaches: insufficient language skills in German or French; pregnancy, lactation, any contraindication for MRI (active implants, passive ferromagnetic implants, passive non-ferromagnetic metallic implants >4cm in the region covered by the active RF coils, large tattoos inside a region covered by the active radiofrequency (RF) coils, claustrophobia or suspected/known non-compliance), smoking within the last 10 years prior recruitment, any other drug consumption except moderate alcohol intake (less than a standard drink containing 10 grams of alcohol per day) or use of medical cannabis, any previous head trauma (with known/suspected intracranial consequences), Body Mass Index (BMI) >30, and any other chronic progressive disease.

  * Specific Criteria for group 1: The calculated biological age (BioAge R Package algorithm) differs by > +/- 3 years from the chronological age. These patients will not be further invited for a study visit with clinical examination and MRI.
  * Specific Criteria for group 2: EDSS > 6.0 as this impacts physical testing; clinical relapse within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: recruitment from the general population through advertisement Group 2: recruitment primarily from the outpatient MS consultation in Inselspital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Brain Age Gap in patients with MS | Up to 2 months after recruitment or finalization of MRI-visit, whichever came first.
  Difference between estimated brain age and (A) biological as well as (B) chronological age.

SECONDARY OUTCOMES:
Relationship of brain age gaps with disease severity | Up to 2 months after recruitment or finalization of MRI-visit, whichever came first.
  Relationship of brain age gaps with disease severity as measured by the expanded disability and severity scale (EDSS; min.-max. according to eligibility criteria: 0-6 points, with a higher score meaning a higher degree of disease severity)
Relationship of brain age gaps with gait speed | Up to 2 months after recruitment or finalization of MRI-visit, whichever came first.
  Relationship of brain age gaps with gait speed as measured by the 25-foot walking test
Relationship of brain age gaps with upper extremity function | Up to 2 months after recruitment or finalization of MRI-visit, whichever came first.
  Relationship of brain age gaps with upper extremity function as measured by the 9-hole Peg Test
Relationship of brain age gaps with sitting-to-raise time | Up to 2 months after recruitment or finalization of MRI-visit, whichever came first.
  Relationship of brain age gaps with a raising test using the sitting-to-raise time
Relationship of brain age gaps with cognitive symptoms | Up to 2 months after recruitment or finalization of MRI-visit, whichever came first.
  Relationship of brain age gaps with cognitive (brief international cognitive assessment in multiple sclerosis (BICAMS))
Relationship of brain age gaps with depression symptoms | Up to 2 months after recruitment or finalization of MRI-visit, whichever came first.
  Relationship of brain age gaps with depression symptoms as assessed with the brief depression inventory (BDI)
Relationship of brain age gaps with fatigue | Up to 2 months after recruitment or finalization of MRI-visit, whichever came first.
  Relationship of brain age gaps with fatigue as assessed with the fatigue severity score (FSS)
Relationship of brain age gaps with quality of life | Up to 2 months after recruitment or finalization of MRI-visit, whichever came first.
  Relationship of brain age gaps with experienced quality of life as assessed with the Multiple Sclerosis Impact Scale (MSIS)-29

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hoepner, PD Dr.med., Principal Investigator — Head of the MS outpatient clinic
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participants data that underlie results in a publication, after deidentification
Supporting Information: Study Protocol
Time Frame: Starting 9 months and ending 48 months after publication
Access Criteria: Encoded data will be provided only to investigators who provide a methodologically sound proposal to achieve the aims in the approved proposal.
  Proposals should be directed to brainage@ikmail.com. To gain access, data requestors will need to sign a data access agreement.
URL: https://clinicaltrials.gov

REFERENCES:
- [Background] Piredda GF, Caneschi S, Hilbert T, Bonanno G, Joseph A, Egger K, Peter J, Kloppel S, Jehli E, Grieder M, Slotboom J, Seiffge D, Goeldlin M, Hoepner R, Willems T, Vulliemoz S, Seeck M, Venkategowda PB, Corredor Jerez RA, Marechal B, Thiran JP, Wiest R, Kober T, Radojewski P. Submillimeter T1 atlas for subject-specific abnormality detection at 7T. Magn Reson Med. 2023 Apr;89(4):1601-1616. doi: 10.1002/mrm.29540. Epub 2022 Dec 7. PMID 36478417
- [Background] Mennecke A, Khakzar KM, German A, Herz K, Fabian MS, Liebert A, Blumcke I, Kasper BS, Nagel AM, Laun FB, Schmidt M, Winkler J, Dorfler A, Zaiss M. 7 tricks for 7 T CEST: Improving the reproducibility of multipool evaluation provides insights into the effects of age and the early stages of Parkinson's disease. NMR Biomed. 2023 Jun;36(6):e4717. doi: 10.1002/nbm.4717. Epub 2022 Mar 17. PMID 35194865
- [Background] Kwon D, Belsky DW. A toolkit for quantification of biological age from blood chemistry and organ function test data: BioAge. Geroscience. 2021 Dec;43(6):2795-2808. doi: 10.1007/s11357-021-00480-5. Epub 2021 Nov 2. PMID 34725754